ExeHeart-Improved Cardiovascular Health for Patients with Inflammatory Joint Diseases: Statistical Analysis Plan (SAP) 2.0

NCT04922840

**Date: March 8th, 2023** 

| Section 1: Administrative information | Index | Description |
|---|---|---|
| Title and trial registration | 1a | ExeHeart- Improved Cardiovascular Health for Patients with Inflammatory Joint Disease: Statistical Analysis Plan |
| | 1b | ClinicalTrials.gov id: NCT04922840 |
| | | REK south-east id: 201227 |
| SAP version | 2 | Data Protection Officer at Diakonhjemmet Hospital id: 00397<br>SAP version 2.0; March 8 <sup>th</sup> , 2023, minor changes to |
| SAI VEISIOII | | SAP version 2.0, March 8 <sup>th</sup> , 2023, minor changes to SAP version 1.0 (29 <sup>th</sup> September, 2022) |
| Protocol version | 3 | https://doi.org/10.1136/bmjopen-2021-058634 |
| SAP revisions | 4a<br>4b | SAP version 2.0 is the first revision of SAP 1.0 |
| | 10 | Amendments in the current version are minor changes from the previous version of SAP: - Items 27a (Analysis methods): VO <sub>2peak</sub> was erroneously stated as covariate in analyses of secondary outcomes. Correct covariate is baseline data of dependent variable. |
| | | - Gender was used as stratification factor in the randomization, but omitted as covariate in ANCOVA |
| | | analyses. This has been remedied in the current version; gender is included as covariate in ANVOCA analyses in addition to age and baseline data of the variable under |
| | | scrutiny. - Post hoc analysis of proportion of patients per group |
| | | acquiring an increase $\ge 3.5 \text{ ml/kg/min}$ at follow-up time |
| | | points (item 27f). This analysis was left out in previous SAP version. |
| | | - Typo < changed to ≥ in item 8: Alternative hypotheses |
| | 4c | Changes in the current version were made at the outset of analyses of longitudinal data from the ExeHeart trial |
| Roles and responsibility | 5 | Anne Therese Tveter; project leader (draft of SAP, critical revision and final approval) Kristine Røren Nordén; PhD student (draft of SAP, critical revision and final approval) Joseph Sexton, statistician (SAP critical revision and final approval) Hanne Dagfinrud, co-supervisor (SAP critical revision and final approval) |
| | | Anne Grete Semb, co-supervisor (SAP critical revision and final approval) |
| | | Jonny Hisdal, co-supervisor (SAP critical revision and final approval) |
| Signatures | 6a | Hutine Rozen Nordin Person writing the SAP (KRN) |
| | 6b | Person writing the SAP (KRN) Senior statistician (IS) |
| | | Senior statistician (JS) |
| | 6c | Anne Therese Tveter |
| | | Anne Therese Neter Chief investigator (ATT) |
| Section 2: Introduction | Index | Description (111) |
| Background and rationale | 7 | Inflammatory joint diseases (IJD), including rheumatoid arthritis (RA), spondyloarthropathy (SpA) and psoriatic arthritis (PsA) are inflammatory autoimmune diseases with common symptoms of joint inflammation, pain, stiffness and fatigue. Compared to the general population, this large patient-group has an increased risk of cardiovascular disease (CVD) and CVD-related mortality. The elevated CVD risk in IJD is only partly attributed to a higher prevalence and burden of traditional risk factors, and the systemic, chronic inflammation is recognized as an independent CVD risk factor. |

Physical activity is inversely associated with risk of metabolic disease, but cardiorespiratory fitness (CRF) has emerged as an even stronger mediator of health outcomes. National and international data show a strong correlation between high levels of CRF and lower risk of CVD and all-cause mortality. In patients with IJD, disease-related factors and uncertainty regarding the dosage of exercise programs are consistent barriers to physical activity. Less time spent at spent at activities with moderate and vigorous intensity may negatively affect CRF and low levels of CRF are reported in patients with IJD. Collectively, the burden of disease and consequent inactivity may be a catalyst for reduced CRF and thus a component of the elevated CVD risk in IJD.

A common notion that intensive exercise can increase disease activity and result in joint destruction and physical discomfort in patients with IJD has previously prevailed, but recent studies demonstrate that vigorous exercise is safe and well-tolerated. High-intensity training (HIIT) is proven superior to exercise at lower intensities in eliciting physiological adaptations. The evidence of HIIT is largely based on supervised clinical trial settings and application of HIIT to real world contexts requires more investigation. Common reservations regarding feasibility, adherence and safety need to be addressed.

Although CRF is identified as a robust physiological marker and a prominent/major risk factor for CVD, assessment of CRF is not included in CVD risk models. A routine measure of CRF as a key vital sign is strongly recommended, though seldom performed in health care settings. CRF is often quantified as peak or maximal oxygen uptake (VO $_{2peak}$ ) and the gold standard for measurement of VO $_{2peak}$  is a CardioPulmonary Exercise Test (CPET). In absence of CPET, non-exercise algorithms that predict VO $_{2peak}$  are viable options. These models use commonly measured clinical variables to estimate CRF and are thereby feasible for use in both primary and specialized clinical care. Notably, the ability of non-exercise algorithms to detect longitudinal change in VO $_{2peak}$  is unclear and presents an important knowledge need.

Objectives

8

Primary aim of the ExeHeart trial is to determine the effect of a 12-week HIIT program set in physiotherapy primary care on CRF in patients with IJD. *Null hypothesis*:

There is no clinically relevant (<3.5 ml/kg/min) between-group difference in change in  $VO_{2peak}$  at 3-month follow-up Alternative hypothesis:

There is a clinically relevant ( $\geq 3.5$  ml/kg/min) between-group difference in change in  $VO_{2peak}$  at 3-month follow-up

Secondary aims are to

a) Assess the long-term effect of a 12-week HIIT program set in physiotherapy primary care on CRF in patients with IJD. *Null hypothesis:* 

There is no clinically relevant (<3.5 ml/kg/min) between-group difference in change in  $VO_{2peak}$  at 6-month follow-up Alternative hypothesis:

There is a clinically relevant ( $\geq 3.5$  ml/kg/min) between-group difference in change in  $VO_{2peak}$  at 6-month follow-up

| | | b) Assess the effect of HIIT on CVD risk factors (blood pressure, cholesterol levels, arterial stiffness, body composition) and disease activity in patients with IJD Null hypotheses: There is no between-group difference in CVD risk factors (blood pressure, cholesterol levels, arterial stiffness, body composition) and disease activity at 3- month follow-up. There is no between-group difference in CVD risk factors (blood pressure, cholesterol levels, arterial stiffness, body composition) and disease activity at 6- month follow-up. Alternative hypotheses: There is a between-group difference in CVD risk factors (blood pressure, cholesterol levels, arterial stiffness, body composition) and disease activity at 3- month follow-up. There is a between-group difference in CVD risk factors (blood pressure, cholesterol levels, arterial stiffness, body composition) and disease activity at 6- month follow-up. c) Assess the association between CRF and disease-specific and CVD-related variables in patients with IJD Null hypothesis: There is no association between CRF and disease-specific and CVD-related variables in patients with IJD Alternative hypothesis: There is one or more associations between CRF and disease-specific and CVD-related variables in patients with IJD d) Explore the feasibility of a HIIT intervention set in physiotherapy primary care is not feasible for patients with IJD in terms of patient's adherence and acceptability Alternative hypothesis: The HIIT intervention set in physiotherapy primary care is deemed feasible for patients with IJD in terms of patient's adherence and acceptability Alternative hypothesis: Patients with IJD in terms of patient's adherence and acceptability Alternative hypothesis: CRF algorithms cannot detect longitudinal change in CRF in patients with IJD Alternative hypothesis: CCRF algorithms can detect longitudinal change in CRF in patients with IJD |
|---|---|---|
| Section 3: Methods | Index | Description |
| Trial design | 9 | Parallel group, randomized controlled trial with repeated measures. Patients are randomly allocated to current clinical practice including CVD risk evaluation, lifestyle advice given at baseline and relevant cardioprotective medication (control group) or current clinical practice and a 12-week HIIT intervention (HIIT group) |
| Randomization | 10 | Study participants are allocated 1:1 by a computer-generated randomization list using permuted blocks of random sizes 4 and 6, stratified by gender. |
| Sample size | 11 | A sample size of 25 in each group will have 80% power to detect a 3.5 mL/kg/min difference in means assuming a reported upper |

| | | bound of standard deviation 4.5 ml/kg/min and a 0.05 two-sided |
|---|---|---|
| | | significance level. Allowing for a possible 20% attrition rate, we will need 60 patients in total, i.e. 30 in each group. |
| Framework | 12 | Superiority trial comparing the effect of HIIT to control |
| Statistical interim analyses and | 13 | The trial will be paused in the case of a serious adverse event |
| stopping guidance | 13 | such as cardiac arrest or death amongst study participants. |
| Timing of final analyses | 14 | Baseline data are to be analyzed following completion of study |
| | | enrollment. All outcomes will be analyzed collectively following completion of study visits for all included patients (anticipated primo 2023). |
| Timing of outcome assessments | 15 | Study visits; baseline, 3 months after baseline (±2 weeks) and 6 months after baseline (±2 weeks) |
| Section 4: Statistical principles | Index | Description |
| Confidence intervals and <i>p</i> -values | 16 | All applicable statistical tests will be two-sided and performed with $\alpha$ = 0.05 |
| | 17 | No adjustment for multiple testing will be done. Significance testing with p-values and 95% confidence intervals (CI) will be reported for the intervention effects on the primary outcome variable. 95% CI will be presented for the intervention effects on all secondary outcome variables (1). |
| | 18 | Two-sided 95% confidence intervals will be reported |
| Adherence and protocol deviations | 19a | Adherence to the intervention will be recorded by use of the training diary. Adherence is set to 70% of HIIT sessions (17 out of 24 possible sessions) |
| | 19b | Attendance to HIIT sessions is tallied by use of the training diary. HIIT exercise intensity sessions will be calculated as mean %HRpeak and Borg RPE 6-20 across sessions and participants. Duration will be reported as mean session duration and average time spent in high intensity intervals. |
| | 19c | The first two weeks of the HIIT intervention may be performed at reduced intensity and/or duration. The HIIT intervention may be downscaled or ceased should the participant present with symptoms such as dizziness or angina pectoris. |
| | 19d | Protocol deviations will be summarized by non-attendance, early session termination, exercise intensity, exercise duration and adverse events |
| | 20 | The primary analysis is an intention-to-treat analysis and will include all randomized patients. The per protocol analysis set will include patients that were randomly assigned to HIIT or control, have baseline and at least one post-baseline measurement of the primary outcome variable and comply to an adherence of ≥70% of HIIT sessions (only applicable to intervention group). |
| Section 5: Trial population | Index | Description |
| Screening data | 21 | Enrolment: the number of months recruiting, the number of patients screened, the number of patients recruited, the number of screened patients not recruited, and the reason for non-recruitment. This summary will be provided overall and presented in the CONSORT flow chart in the publication of trial results. Reasons for declining to participate (time constrains, distance to PT clinic, medical issues, satisfied with current exercise regime, other) and failure to meet eligibility criteria (see index #22) will be tallied and reported |
| Eligibility | 22 | Inclusion criteria: • Age 18-70 • BMI 18.5-40 • Able to walk unaided ≥15 minutes • IJD verified by physician • Norwegian or English speaking |

| | | Evolucion anitanis | | |
|---|---|---|---|---|
| | | Exclusion criteria: | 1/ | |
| | | Lower extremity injury | | gery <12 months |
| | | <ul> <li>Primary neurological di</li> </ul> | isease | |
| | | <ul> <li>Cognitive impairment</li> </ul> | | |
| | | • Participation in high-intensity exercise ≥ 1 session/week in the last 3 months | | |
| | | <ul> <li>American College of Sp</li> </ul> | | ` ' |
| | | | contraindication to maximal exercise test | |
| Recruitment | 23 | A CONSORT flow diagram | | ed to summarize the |
| | | number of patients who wer | | _ |
| | | assessed for eligibility a | | |
| | | • ineligible at screening of | or declined | to participate |
| | | • randomized | 1 11 | |
| | | received the randomize | | n |
| | | discontinued the intervent | | |
| | | • did not receive the HII7 | | |
| | | • included in primary and | | nonths |
| | | • lost to follow-up at 3 m | | |
| | | • included in primary and | | nonths |
| W. 1 1 1/0 H | | • lost to follow-up at 6 m | | 0 0 11 |
| Withdrawal/follow-up | 24a | Withdrawal from the interve | | |
| | 2.41 | assessments will be reported | | |
| | 24b+ | The number of losses to foll | | |
| | С | 3-month and 6-month time parm | point will t | be summarized by treatment |
| Baseline patient characteristics | 25a | | mmy tahla | s of baseline |
| Basefine patient characteristics | 234 | Please see table 1 and 2 (dummy tables of baseline characteristics). | | |
| | 25b | Categorical data will be pres | sented as n | umbers (percentages) |
| | 250 | Continuous data will be pres | | |
| | | median (IQR) if skewedly d | | |
| | | The clinical importance of any imbalance between groups will be | | |
| | | discussed, but no tests of sta | itistical sig | nificance will be performed |
| Section 6 Analysis | Index | Description | | |
| Outcome definitions | 26 | Please see protocol article for procedures (2) | or descripti | ion of data collection |
| | | procedures (2) | | |
| | | Primary outcome (unit) | Time | Primary effect estimates |
| | | Peak oxygen uptake (VO <sub>2peak</sub> , | Baseline, | Change from baseline-3mo |
| | | mL·kg-1·min-1 and L·min-1) | 3 mo, 6 | (95% CI) |
| | | Secondary outcomes (unit) | Time | Primary effect estimates |
| | | Spirometry | Baseline, | Change from baseline-3mo |
| | | Forced Vital Capacity (FVC, | 3mo, | (95% CI) |
| | | L) Forced Expiratory Volume | 6mo | |
| | | (FEV1, L) | | |
| | | Peak Expiratory Flow (PEF, | | |
| | | L·min-1) | | |
| | | Maximal Voluntary Ventilation (MVV, L·min <sup>-1</sup> ) | | |
| | | Peak HR (HR <sub>peak</sub> , beat·min <sup>-1</sup> ) | Baseline, | Change from baseline-3mo |
| | | | 3mo,<br>6mo | (95% CI) |
| | | Ventilatory threshold 1 | Baseline, | Change from baseline-3mo |
| | | | 3mo, | (95% CI) |
| | | Ventilatory threshold 2 | 6mo<br>Baseline, | Change from baseline-3mo |
| | | v chiliatory uneshold 2 | 3mo, | (95% CI) |
| | | | 6mo | |
| | 1 | Maximum minute ventilation at | Baseline, | Change from baseline-3mo |
| | | | 3mo | |
| | | peak exercise (V <sub>Emax</sub> , L·min <sup>-1</sup> ) | 3mo,<br>6mo | (95% CI) |

| 6mo | |
|---|---|
| Baseline,<br>3mo,<br>6mo | Change from baseline-3m (95% CI) |
| Baseline,<br>3mo,<br>6mo | Chi-square (or exact test i<br>overall total <40) |
| Baseline,<br>3mo,<br>6mo | Change from baseline-3m (95% CI) |
| Baseline,<br>3mo,<br>6mo | Chi-square (or exact test is overall total <40) |
| | Samo, 6mo Baseline, 3mo, 6mo |

| | | Use of medication; analgesics, IJD and CVD medication | | |
|---|---|---|---|---|
| | | BASFI (for SpA) (0-10) Covid-19 infection and/or | Baseline, | Descriptive per treatment |
| | | quarantine in the past 3 months | 3mo,<br>6mo | arm |
| | | EuroQol-5D-5L (-0.59 to 1) | Baseline,<br>3mo,<br>6mo | Change from baseline-3mo (95% CI) |
| | | EuroQol-5D-5L VAS (0-100) | Baseline,<br>3mo,<br>6mo | Change from baseline-3mo (95% CI) |
| | | Numerical Rating Scale<br>Pain (0-10)<br>Fatigue (0-10) | Baseline,<br>3mo,<br>6mo | Change from baseline-3mo (95% CI) |
| | | Physical activity index (0-45) | Baseline,<br>3mo,<br>6mo | Change from baseline-3mo (95% CI) |
| | | Exercise beliefs and exercise habits (mean 1-5 for each domain) | Baseline,<br>3mo,<br>6mo | Change from baseline-3mo (95% CI) |
| Analysis methods | 27a | Primary outcome: ANCO | | render and VO <sub>2peak</sub> |
| | = / • • | (a) baseline to be included as | | |
| | | Secondary outcomes (please | | |
| | | objectives: | | r · · · |
| | | a) ANCOVA. Age, gende | r and basel | line data of dependent |
| | | variable to be included | as covariat | tes. |
| | | b) ANCOVA. Age, gende | | |
| | | variable to be included | | |
| | | c) Multiple linear regressi | | |
| | | variables as independen | nt variables | s to VO <sub>2peak</sub> (dependent |
| | | variable) | 14 | analonia ta ba danidad in |
| | | <ul> <li>d) Descriptive statistics, exploratory analysis to be decided in light of final data set</li> <li>e) Evaluated by correlation, illustrated with Bland-Altman plot Table 3 is a dummy table on the effect of the HIIT intervention or cardiorespiratory and cardiovascular variables at 3-month follow-</li> </ul> | | |
| | | up. Table 4 is a dummy table on the effect of the HIIT | | |
| | | intervention on PROMS and disease-related variables at 3-month | | |
| | | follow-up. | | |
| | 27b | Age, VO <sub>2peak</sub> values at baseline and other relevant factors such as | | |
| | ļ | IJD entity | | |
| | 27c | Primary outcome: | | . 110 |
| | | ANCOVA; dependent varia | | |
| | | continuous variable with no | | , <del>-</del> |
| | | VO <sub>2peak</sub> at baseline) are concategorical variable (group | | |
| | | stratification factor and furt | | |
| | | The following assumptions | | |
| | | variance (Levene's test), ske | | |
| | | relationships. | | |
| | 27d | Regarding ANCOVA; variable transformation will be consider in case of violations. | | |
| | | Dorometric and non never- | trio statisti | ool analysees will be seemied |
| | | Parametric and non-parame out as appropriate based on | | |
| | | distribution (q-q plots and h | | |
| | | regarding the normal probal univariate normality will be | bility curve | |
| | 27e | Sensitivity analyses of prim violations of analysis assum | ary outcon | |
| | 250 | of skewed residuals | | |
| | 27f | Subgroup analysis of per-pr | otocol pop | ulation in HIIT group |

| Missing data 28 Sensitivity analyses with different methods for handling missing data such as; - Complete case analysis - Single imputation such as last observation carried forward of simple mean imputation - Multiple imputation Additional analyses 29 Per protocol (as defined by index #20) of primary and secondary outcome variables All adverse event (AE) and serious adverse events (SAE) are recorded in a data file and the following information is described. • AE or SAE • Severity; mild (cold/flu), moderate (requires medical attention), serious (hospitalization, malignant disease, death start and end data of event • Study causality; no/possibly/yes • Patient consequence • Trial consequence • Trial consequence • Trial consequence SAE will be reported to the project leader, who in turn will decident on further study participation and referral to relevant physician such as GP, rheumatologist, cardiologist. All events will be coded, categorized and summarized. The number and percentage of AE and SAE will be reported per treatment arm. No formal statistical testing. Statistical software 31 STATA 16.1 References 32a No plan to include nonstandard statistical methods Patient questionnaires: Encrypted data will be sent from nettskjema, no to Sensitive Data Services (TSD) at the Universit of Oslo, and downloaded to secure research server at Diakonhjemmet Hospital. Patients case report forms: Secured in locked cabinets according to hospital policy and remain stored for 5 years after study completion. All data files will be stored on the secure research server at Diakonhjemmet Hospital with access to files restricted to the following project group members KRN, HD, AGS, JSe, CF, EB and ATT. 32c N/Forskning/ExeHeart/Data/DataExeHeart.xls Guidelines for the Content of Statistical Analysis Plans in Clinical Trials (3) | | | Post hoc analyses of proportion of patients per group with an |
|---|---|---|---|
| Additional analyses 29 Per protocol (as defined by index #20) of primary and secondary outcome variables All adverse event (AE) and serious adverse events (SAE) are recorded in a data file and the following information is described. AE or SAE Severity; mild (cold/flu), moderate (requires medical attention), serious (hospitalization, malignant disease, death Start and end data of event Study causality; no/possibly/yes Patient consequence Trial consequence SAE will be reported to the project leader, who in turn will decident on further study participation and referral to relevant physician such as GP, rheumatologist, cardiologist. All events will be coded, categorized and summarized. The number and percentage of AE and SAE will be reported per treatment arm. No formal statistical testing. Statistical software 31 STATA 16.1 References 32a No plan to include nonstandard statistical methods Patient questionnaires: Encrypted data will be sent from nettskjema.no to Sensitive Data Services (TSD) at the Universit of Oslo, and downloaded to secure research server at Diakonhjemmet Hospital. Patients case report forms: Secured in locked cabinets according to hospital policy and remain stored for 5 years after study completion. All data files will be stored on the secure research server at Diakonhjemmet Hospital with access to files restricted to the following project group members KRN, HD, AGS, JSe, CF, EB and ATT. 32c N/Forskning/ExeHeart/Data/DataExeHeart.xls Guidelines for the Content of Statistical Analysis Plans in Clinical Trials (3) | Missing data | 28 | <ul> <li>Complete case analysis</li> <li>Single imputation such as last observation carried forward or simple mean imputation</li> </ul> |
| recorded in a data file and the following information is described. AE or SAE Severity; mild (cold/flu), moderate (requires medical attention), serious (hospitalization, malignant disease, death Start and end data of event Study causality; no/possibly/yes Patient consequence Trial consequence SAE will be reported to the project leader, who in turn will decion further study participation and referral to relevant physician such as GP, rheumatologist, cardiologist. All events will be coded, categorized and summarized. The number and percentage of AE and SAE will be reported per treatment arm. No formal statistical testing. Statistical software 31 STATA 16.1 References 32a No plan to include nonstandard statistical methods Patient questionnaires: Encrypted data will be sent from nettskjema.no to Sensitive Data Services (TSD) at the Universit of Oslo, and downloaded to secure research server at Diakonhjemmet Hospital. Patients case report forms: Secured in locked cabinets according to hospital policy and remain stored for 5 years after study completion. All data files will be stored on the secure research server at Diakonhjemmet Hospital with access to files restricted to the following project group members KRN, HD, AGS, JSe, CF, EB and ATT. 32c N/Forskning/ExeHeart/Data/DataExeHeart.xls Guidelines for the Content of Statistical Analysis Plans in Clinical Trials (3) | Additional analyses | 29 | Per protocol (as defined by index #20) of primary and secondary |
| References 32a No plan to include nonstandard statistical methods 32b Patient questionnaires: Encrypted data will be sent from nettskjema.no to Sensitive Data Services (TSD) at the Universit of Oslo, and downloaded to secure research server at Diakonhjemmet Hospital. Patients case report forms: Secured in locked cabinets according to hospital policy and remain stored for 5 years after study completion. All data files will be stored on the secure research server at Diakonhjemmet Hospital with access to files restricted to the following project group members KRN, HD, AGS, JSe, CF, EB and ATT. 32c N/Forskning/ExeHeart/Data/DataExeHeart.xls 32d Guidelines for the Content of Statistical Analysis Plans in Clinical Trials (3) | Harms/adverse events | 30 | <ul> <li>All adverse event (AE) and serious adverse events (SAE) are recorded in a data file and the following information is described;</li> <li>AE or SAE</li> <li>Severity; mild (cold/flu), moderate (requires medical attention), serious (hospitalization, malignant disease, death)</li> <li>Start and end data of event</li> <li>Study causality; no/possibly/yes</li> <li>Patient consequence</li> <li>Trial consequence</li> <li>SAE will be reported to the project leader, who in turn will decide on further study participation and referral to relevant physician such as GP, rheumatologist, cardiologist.</li> <li>All events will be coded, categorized and summarized. The number and percentage of AE and SAE will be reported per</li> </ul> |
| Patient questionnaires: Encrypted data will be sent from nettskjema.no to Sensitive Data Services (TSD) at the Universit of Oslo, and downloaded to secure research server at Diakonhjemmet Hospital. Patients case report forms: Secured ir locked cabinets according to hospital policy and remain stored for 5 years after study completion. All data files will be stored on the secure research server at Diakonhjemmet Hospital with access to files restricted to the following project group members KRN, HD, AGS, JSe, CF, EB and ATT. 32c N/Forskning/ExeHeart/Data/DataExeHeart.xls Guidelines for the Content of Statistical Analysis Plans in Clinical Trials (3) | | | |
| Guidelines for the Content of Statistical Analysis Plans in Clinical Trials (3) | References | 32b | Patient questionnaires: Encrypted data will be sent from nettskjema.no to Sensitive Data Services (TSD) at the University of Oslo, and downloaded to secure research server at Diakonhjemmet Hospital. Patients case report forms: Secured in locked cabinets according to hospital policy and remain stored for 5 years after study completion. All data files will be stored on the secure research server at Diakonhjemmet Hospital with access to files restricted to the following project group members KRN, HD, AGS, JSe, CF, EB and ATT. |
| T II 1 (A) | | | Guidelines for the Content of Statistical Analysis Plans |

Table 2: Dummy table of baseline characteristics. Data are presented as mean (SD) unless otherwise indicated.

| Total<br>N= | HIIT group<br>N= | Control group<br>N= |
|-------------|------------------|---------------------|

ACE inhibitors: angiotensin-converting enzyme inhibitor, CRP: C-reactive protein, CVD: cardiovascular disease, DMARDs: disease-modifying anti-rheumatic drugs, ESR: erythrocyte sedimentation rate, HDL: high-density lipoprotein, JAKi: Janus Kinase inhibitors, LDL: low-density lipoprotein, NSAIDs: non-steroidal anti-inflammatory drugs, RA: rheumatoid arthritis, PsA: psoriatic arthritis, SCORE2: Systemic COronary Risk Estimation 2, SpA: spondyloarthritis

Table 3: Dummy table of baseline characteristics (supplementary files). Data are presented as mean (SD) unless otherwise indicated.

| Baseline characteristics | Total | HIIT group | Control group |
|---------------------------------------|-------|------------|---------------|
| CPET variables | N= | N= | N= |
| Forced vital capacity, L | | | |
| Forced expiratory volume, L | | | |
| Peak expiratory flow, L/min | | | |
| Maximal voluntary ventilation, L/min | | | |
| VT1 | | | |
| VO <sub>2</sub> mL/kg/min | | | |
| HR | | | |
| VT2 | | | |
| VO <sub>2</sub> mL/kg/min | | | |
| HR | | | |
| Breathing reserve at peak exercise, % | | | |
| $VE/VO_2$ | | | |
| at VT1 | | | |
| at VT2 | | | |
| VE/VCO <sub>2</sub> | | | |
| at VT1 | | | |
| atVT2 | | | |
| Clinical disease activity | | | |
| DAS28 | | | |
| DAPSA | | | |
| ASDAS | | | |
| D : : (0) | | | |
| Remission, n (%) | | | |
| Low, n (%) | | | |
| Moderate, n (%) | | | |
| High, n (%) | | | |
| Self-reported disease activity | | | |
| RAID, 0-10, 10= worst | | | |
| PsAID, 0-10, 10= worst | | | |
| BASDAI, $0-10$ , $10=$ severe | | | |
| BASFI, 0-10, 10= impossible | | | |
| BAS-G, 0-10, 10= very severe | | | |

ASDAS: Ankylosing Spondylitis Disease Activity Score, BASDAI: Bath Ankylosing Spondylitis Disease Activity Index, BASFI: Bath Ankylosing Spondylitis Functional Index, BAS-G: Bath Ankylosing Spondylitis Patient Global Score, CPET: cardiopulmonary exercise test, DAS28: Disease Activity Score Calculator for RA, DAPSA: Disease Activity Index for PSoriatic Arthritis, HR: heart rate, RAID: Rheumatoid Arthritis Impact of Disease, PsAID: Psoriatic Arthritis Impact of Disease, VCO<sub>2</sub>: volume of carbon dioxide, V<sub>E</sub>: minute ventilation, VO<sub>2</sub>: volume of oxygen, VT1: ventilatory threshold 1, VT2: ventilatory threshold 2

Table 4: Dummy table of effect of HIIT on cardiorespiratory fitness and other cardiovascular disease risk factors at 3-month follow-up. Data are presented as mean (SD) unless otherwise indicated.

| | HII | T group | Con | trol group | Mean group<br>difference<br>(95%CI) |
|---|---|---|---|---|---|
| | Baseline | 3 months | Baseline | 3 months | |
| Cardiorespiratory fitness | | | | | |
| VO <sub>2peak</sub> , ml/kg/min | | | | | |
| VO <sub>2peak</sub> , L/min | | | | | |
| VO <sub>2peak</sub> , ml/FFM | | | | | |
| Peak HR | | | | | |
| RER | | | | | |
| V <sub>E</sub> at peak exercise | | | | | |
| Borg RPE 0-10, 10= max | | | | | |
| Lactate, mmol/L | | | | | |
| Resting HR, beat/min | | | | | |
| Lipids | | | | | |
| Total cholesterol, mmol/L | | | | | |
| HDL, mmol/L | | | | | |
| LDL, mmol/L | | | | | |
| Triglycerides, mmol/L | | | | | |
| Blood pressure | | | | | |
| Systolic, mm Hg | | | | | |
| Diastolic, mm Hg | | | | | |
| Mean arterial pressure, mm Hg | | | | | |
| SCORE2 | | | | | |
| Arterial stiffness | | | | | |
| Augmentation index | | | | | |
| Pulse wave velocity, m/s | | | | | |
| Anthropometric measures | | | | | |
| BMI, kg/m <sup>2</sup> | | | | | |
| Waist circumference, cm | | | | | |
| Fat mass, kg | | | | | |
| Fat-free mass, kg | | | | | |
| Visceral fat indicator | | | | | |

Borg RPE: Borg rating of perceived exertion, BMI: body mass index, FFM: fat-free mass, HDL: high-density lipoprotein, HR: heart rate, LDL: low-density lipoprotein, RER: respiratory exchange ratio, SCORE2: Systemic COronary Risk Estimation 2, V<sub>E</sub>: minute ventilation, VO<sub>2peak</sub>: peak oxygen uptake,

Table 5: Dummy table of effect of HIIT on disease activity and patient-reported outcomes at 3-month follow-up. Data are presented as mean (SD) unless otherwise indicated.

| | нит | f group | Conti | ol group | Mean group<br>difference<br>(95%CI) |
|---|---|---|---|---|---|
| | Baseline | 3 months | Baseline | 3 months | |
| Clinical disease activity | | | | | |
| Remission, n (%) | | | | | |
| Low, n (%) | | | | | |
| Moderate, n (%) | | | | | |
| High, n (%) | | | | | |
| Inflammatory markers | | | | | |
| CRP, mg/L | | | | | |
| ESR, mm | | | | | |
| Self-reported measures of disease | | | | | |
| activity and health | | | | | |
| RAID, 0-10, 10=worst | | | | | |
| PsAID, 0-10, 10=worst | | | | | |
| BASDAI, 0-10, 10=severe | | | | | |
| BASFI, 0-10, 10= impossible | | | | | |
| BAS-G, 0-10, 10= very severe | | | | | |
| NRS Pain last week, 0-10, 0= no pain | | | | | |
| NRS Fatigue last week, 0-10, 0= no | | | | | |
| fatigue | | | | | |
| EuroQol-5D-5L utility index, 0-1, 1= best | | | | | |
| health state | | | | | |
| EuroQol-5D-5L, VAS 0-100, 100= best | | | | | |
| imaginable health | | | | | |
| Exercise beliefs | | | | | |
| Self-efficacy | | | | | |

| Barriers to exercise |
|---------------------------|
| Benefits of exercise |
| Impact of exercise on IJD |
| Physical activity index |

BASDAI: Bath Ankylosing Spondylitis Disease Activity Index, BASFI: Bath Ankylosing Spondylitis Functional Index, BAS-G: Bath Ankylosing Spondylitis Patient Global Score, CRP: C-reactive protein, ESR: erythrocyte sedimentation rate, NRS: Numeric rating scale, RAID: Rheumatoid Arthritis Impact of Disease, PsAID: Psoriatic Arthritis Impact of Disease,

## **References:**

- 1. Harrington D, D'Agostino RB, Sr., Gatsonis C, Hogan JW, Hunter DJ, Normand ST, et al. New Guidelines for Statistical Reporting in the Journal. The New England journal of medicine. 2019;381(3):285-6.
- 2. Nordén KR, Dagfinrud H, Semb AG, Hisdal J, Viktil KK, Sexton J, et al. Effect of high-intensity exercise on cardiorespiratory fitness, cardiovascular disease risk and disease activity in patients with inflammatory joint disease: protocol for the ExeHeart randomised controlled trial. BMJ open. 2022;12(2):e058634.
- 3. Gamble C, Krishan A, Stocken D, Lewis S, Juszczak E, Doré C, et al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. Jama. 2017;318(23):2337-43.